CLINICAL TRIAL: NCT00743925
Title: FRANCIS-ACS Trial: A Study of the Safety and Efficacy of A 002 in Subjects With Acute Coronary Syndromes
Acronym: FRANCIS-ACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN-CVD2224
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-01

CONDITIONS: Acute Coronary Syndrome
Keywords: Unstable Angina; STEMI; NSTEMI; ACS; Acute Coronary Syndrome; C14.280.647.124; C14.280.647.500
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction | interventions — varespladib methyl; varespladib; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): A-002 (500 mg QD) plus Atorvastatin (80 mg QD)
  Interventions: Drug: Varespladib Methyl (A-002)
- 2 (Placebo Comparator): Matching Placebo tablets plus Atorvastatin (80 mg QD)
  Interventions: Drug: Varespladib Methyl (A-002)

INTERVENTIONS:
Drug: Varespladib Methyl (A-002) — 2 Tablets (250 mg each) once daily for at least 24 weeks in combination with Atorvastatin (80 mg tablet once a day).
  Other Names: A-002; Varespladib; Lipitor; Atorvastatin

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of A 002 when added to high dose atorvastatin in subjects with an acute coronary syndrome (ACS)

DETAILED DESCRIPTION:
This is a double-blind randomized parallel group placebo controlled study in subjects presenting with an ACS. Subjects will be randomized to receive either A 002 500 mg once daily (QD) or placebo tablets in addition to 80 mg atorvastatin QD.

Randomization must occur within ≤96 hours of hospital admission for the index ACS event, or, if already hospitalized, within ≤96 hours of index event diagnosis. Follow-up visits will occur at Weeks 2, 4, 8, 12, 16, 20, and 24 post-randomization; and monthly thereafter until study completion.

All enrolled subjects will remain on treatment until all subjects have been treated for a minimum of 24 weeks or until the occurrence of a Major Adverse Cardiac Event (MACE). At that point, all active subjects (those who have not early withdrawn or those that have not already had a MACE) will be brought in for a Final Study Visit. Subjects who complete the Final Study Visit may be eligible to enroll in an open-label extension study for up to 2 years total study drug exposure.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥18 years of age
* A diagnosis of unstable angina, NSTEMI, or STEMI
* Any one of the following criteria: Diabetes, CRP ≥2 mg/L, or metabolic syndrome
* Subjects must be randomized within 96 hours of the index event
* Percutaneous revascularization, if required or planned, must occur prior to randomization

Exclusion Criteria:

- Subjects must NOT meet any of the following exclusion criteria:

* Subjects enrolled in another experimental (interventional) protocol within the past 30 days prior to Screening.
* Subjects treated for cancer within the previous 5 years except for skin basal cell carcinoma or carcinoma in situ of the cervix, with measures other than a minor, complete surgical excision (e.g., chemotherapy), or radiation therapy.
* The presence of severe liver disease with cirrhosis, recent active hepatitis, active chronic hepatitis, ALT or AST >3 x ULN, biliary obstruction with hyperbilirubinemia (total bilirubin >2 x ULN)
* Active cholecystitis, gall bladder symptoms, or potential hepato-biliary abnormalities
* The presence of severe renal impairment (CrCl <30 mL/min or creatinine >3 x ULN), nephrotic syndrome, or patients undergoing dialysis
* Uncontrolled diabetes mellitus (HbA1c >11% within the last 1 month prior to Screening)
* Females who are nursing, pregnant, or intend to become pregnant during the time of the study, or females of child-bearing potential who have a positive pregnancy test during screening evaluation. Women of child-bearing potential must also use a reliable method of birth control during the study and for 1 month following completion of therapy. A reliable method for this study is defined as one of the following: oral or injectable contraceptives, IUD, contraceptive implants, tubal ligation, hysterectomy, a barrier method (diaphragm with spermicidal foam or jelly, or a condom).
* Subjects who have a history of alcohol or drug abuse within 1 year of study entry
* Subjects living too far from participating center or unable to return for follow-up visits
* Subjects who in the opinion of the Investigator are a poor medical or psychiatric risk for therapy with an investigational drug, are unreliable, or have an incomplete understanding of the study which may affect their ability to take drugs as prescribed or comply with instructions
* Known HIV, Hepatitis B or C virus, or tuberculosis infection
* Acute bacterial, fungal or viral infection
* Any current statin therapy at maximum recommended dosage. For atorvastatin, fluvastatin, lovastatin, pravastatin and simvastatin 80 mg QD at the time of the index event and for rosuvastatin 20 mg QD to 40 mg QD
* Drugs that are potent inhibitors of cytochrome P450 unless they can be withdrawn
* Subjects with NYHA Class III or IV heart failure, or LVEF <30
* Subjects with moderate or severe aortic stenosis, aortic regurgitation, mitral stenosis or mitral regurgitation
* Ventricular arrhythmias requiring chronic drug treatment or ICD
* Subjects with no stenosis or stenosis <50% on angiography
* Subjects with a pacemaker or persistent LBBB
* LDL-C >200 mg/dL (5.2 mmol/L)
* Fasting triglyceride levels of ≥400 mg/dL (4.5 mmol/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 625 (Actual)
Dates: Start 2008-07; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Mean percent changes in LDL hs-CRP, sPLA2 and other biomarkers will be compared between the 2 treatment groups. | 8 Weeks

SECONDARY OUTCOMES:
The occurrence of MACEs will be examined for any treatment-related trends at study completion. | End of Study

CONTACTS AND LOCATIONS:
Locations (41):
- Georgia (10):
  - Cardiological hospital of The Patriarchate of all Georgia, Tbilisi
  - Tbilisi State Medical University, Al. Aladashvili University Clinic, Tbilisi
  - Cardio Reanimation Centre, Tbilisi
  - Cardiological Clinic "Guli", Tbilisi
  - Tbilisi LTD Cardiology Clinic, Tbilisi
  - Emergency Cardiology Center by acad. G. Chapidze, Tbilisi
  - National Center of Therapy, Tbilisi
  - Multiprofile Clinical Hospital of Tbilisi #2, Tbilisi
  - Diagnostic Services Clinic, Tbilisi
  - Limited Company "ADAPTI" The Clinic of Angiocardiology "ADAPTI", Tbilisi
- Russia (20):
  - Municipal Healthcare Institution, Gatchina
  - Municipal Healthcare Institution, Kemerovo
  - Non-State Healthcare Institution, Kemerovo
  - Krasnoyarsk Medical Academy, Krasnoyarsk
  - State Healthcare Intstitution of Moscow, Moscow
  - City Clinical Hospital №12, Nizhny Novgorod
  - Municipal Healthcare Institution, Novosibirsk
  - Regional State Healthcare Institution, Novosibirsk
  - Municipal Healthcare Institution, Perm
  - St.Petersburg State Healthcare Institution, Saint Petersburg
  - State Educational Institution for Further Professional Training, Saint Petersburg
  - Federal State Healthcare Institution, Saint Petersburg
  - State Healthcare Institution, Saint Petersburg
  - Saint-Petersburg State Healthcare Institution, Saint Petersburg
  - State Healthcare Institution, Samara
  - Saratov State Medical University, Saratov
  - Federal State Institution, Saratov
  - State Institution Research Cardiology Institute, Tomsk
  - Tyumen Cardiology Center,, Tyumen
  - New Hospital Medical Union, Yekaterinburg
- Ukraine (11):
  - Municipal Clinical Hospital No. 27, Kharkiv
  - Department of Cardiology of Central Clinical Hospital, Kharkiv
  - L.T. Malaya Institute of Therapy of AMS of Ukraine, Kharkiv
  - Kharkiv Medical Academy of Post-Graduate Education, Kharkiv
  - Kyiv City Clinical Hospital #1, Kyiv
  - National Scientific Center, Kyiv
  - Lviv Danylo Halytsky National University, Lviv
  - Lviv Regional State Clinical Treatment and Diagnostics Cardiology Center, Lviv
  - Uzhgorod National University, Uzhhorod
  - Zaporizhzhya Regional Cardiological Dispensary, Zaporizhzhya
  - Zhytomyr city hospital #1, Zhytomyr

REFERENCES:
- [Derived] Rosenson RS, Hislop C, Elliott M, Stasiv Y, Goulder M, Waters D. Effects of varespladib methyl on biomarkers and major cardiovascular events in acute coronary syndrome patients. J Am Coll Cardiol. 2010 Sep 28;56(14):1079-88. doi: 10.1016/j.jacc.2010.06.015. PMID 20863951
- See also: Sponsor's Website — http://www.anthera.com/